CLINICAL TRIAL: NCT05268302
Title: Phase One, Open Label, Assessment of a Dengue-4-Virus-Live Virus Human Challenge - (DENV-4-LVHC) Virus Strain in Healthy U.S. Adults
Brief Title: Dengue 4 Human Infection Model (Dengue CVD 11000; DHIM-4)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Medical Technology Enterprise Consortium (MTEC) (Unknown)
Responsible Party: Principal Investigator, Kirsten Lyke, Principal Investigator, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00087533
Record Dates: First submitted 2022-02-09; First posted 2022-03-07 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Primary (Experimental): 0.95 x 10^2 Plaque Forming Units
  Interventions: Biological: Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Low Dose
- Low Dose Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Homologous Rechallenge (Experimental): 0.95 x 10^2 Plaque Forming Units
  Interventions: Biological: Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Low Dose - Homologous Rechallenge

INTERVENTIONS:
Biological: Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Low Dose — Low dose 0.5 mL of the challenge strain is administered subcutaneously in the triceps region of the arm on Study Day 0.
  Arms: Low Dose Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Primary
Biological: Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Low Dose - Homologous Rechallenge — Low dose 0.5 mL of the challenge strain is administered subcutaneously in the triceps region of the arm on Study Day 366 in previously dosed participants.
  Other Names: Homologous Rechallenge
  Arms: Low Dose Dengue 4 Live Virus Human Challenge (DENV-4-LVHC) - Homologous Rechallenge

SUMMARY:
The purpose of this research study is to test a weakened form of an experimental dengue virus challenge at different doses to test if participants develop symptoms or circulating virus in the blood (called viremia). When volunteers are exposed to dengue on purpose, it is called a "challenge" or Dengue Human Infection Model (DHIM). The research team is collecting information about the safety of the challenge and the best dose to use. The information may help us to make a dengue challenge (a DHIM) that will test vaccines to protect people from dengue.

DETAILED DESCRIPTION:
The purpose of this research study is to test a weakened form of an experimental dengue virus challenge at different doses to test if participants develop symptoms or circulating virus in the blood (called viremia). When volunteers are exposed to dengue on purpose, it is called a "challenge" or Dengue Human Infection Model (DHIM). The research team is collecting information about the safety of the challenge and the best dose to use. The information may help the research team to make a dengue challenge (a DHIM) that will test vaccines to protect people from dengue. The duration of participation will last for 180 days (six months) after challenge including up to 22 visits. After participants are exposed to the weakened dengue virus, the research team will follow them closely to measure their symptoms. Like the flu, participants might expect to have a headache, rash, body aches, fever and chills or they may experience no symptoms whatsoever. If participants do develop symptoms, the research team will monitor them closely in a local hotel or a wing of our hospital to ensure safety and to treat symptoms if they occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breastfeeding female between 18 and 50 years of age (inclusive) at the time of consent
* Volunteers must be able to provide written informed consent.
* Volunteers must be healthy as established by medical history and clinical examination at study entry
* Volunteers must pass a comprehension test and be able to comply with all study requirements.
* Female volunteers of non-childbearing potential (non-childbearing potential is defined as having had one of the following: a tubal ligation at least 3 months prior to enrollment, a hysterectomy, an ovariectomy, or is post-menopausal).
* Female volunteers of childbearing potential may be enrolled in the study, if all the following apply:
* Practiced adequate contraception for 30 days prior to challenge
* Has a negative urine pregnancy test on the day of DHIM
* Agrees to continue adequate contraception until two months after completion of the DHIM

Exclusion Criteria:

* History of dengue infection or dengue illness, or history of flavivirus infection or vaccination (e.g., yellow fever, tick-borne-encephalitis virus [TBEV], Japanese encephalitis, and dengue) (Note: for the homologous rechallenge sub-study, criteria does not apply)
* Volunteers positive for antibodies to flaviviruses (FV) to include dengue virus, West Nile virus, Yellow Fever virus, Zika virus, and Japanese encephalitis virus. (Note: for the homologous rechallenge sub-study, criteria does not apply)
* Planned administration of any flavivirus vaccine for the entire study duration
* Any recent (within 4 weeks) or planned travel to any dengue endemic area while participating in the trial
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required)
* Volunteer seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* Safety laboratory test results at screening that are deemed clinically significant or more than Grade 1 deviation from normal with the exception of PT/PTT, fibrinogen decrease, ALT/AST increase (acceptable to 1.1 ULN), platelet decrease which will be exclusionary at Grade 1 or higher
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* History of bipolar disorder, schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the volunteer from participating in the study
* Significant screening physical examination abnormalities at the discretion of the investigator, including a BMI > 35 kg/m2
* Planned administration or administration of a vaccine/product not planned in the study protocol during the period starting 30 days prior to the DHIM until 56 days after the study completion (routine influenza or COVID-19 vaccination will be allowed if it is not administered within 14 days preceding DHIM)
* Use of any investigational or non-registered product (drug or vaccine) other than the study DHIM during the period starting 30 days preceding the DHIM and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the DHIM (for corticosteroids, this will mean prednisone 5 mg/day or equivalent; inhaled, intranasal and topical steroids are allowed)
* Concurrently participating in another clinical study, at any time during the study period, in which the volunteer has been or will be exposed to an investigational or a noninvestigational product (pharmaceutical product or device)
* Autoimmune disease or history of autoimmune disease
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study product or related to a study procedure
* Major congenital defects or serious chronic illness
* History of any neurological disorders or seizures
* Acute disease and/or fever (≥37.5°C/99.5°F oral body temperature) at the time of enrollment: note that a volunteer with a minor illness such as mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator
* Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the DHIM or planned administration during the study period
* Recent history of chronic alcohol consumption (more than 2 drinks per day and/or drug abuse) based on volunteer reported history
* Pregnant or breastfeeding female or female currently planning to become pregnant or planning to discontinue adequate contraception
* Men who intend to father a child during the study period (approximately 2 months)
* Any religious or personal beliefs that bar the administration of blood products, transfusions or serum albumin
* Planned or current administration of an HMG-CoA reductase inhibitor (i.e., lovastatin, simvastatin, atorvastatin, etc.)
* Currently regularly taking anti-coagulant medication, aspirin, or non-steroidal anti-inflammatory drugs (NSAIDs)
* Any other condition which, in the opinion of the investigator, prevents the volunteer from participating in the study
* Temporary Exclusion Criteria:
* Acute disease and/or fever (> 38°C/100.4°F oral body temperature) at the time or within 6 hours of challenge inoculation: note that a volunteer with a minor illness such as mild upper respiratory infection, etc., without fever, and with a negative SARS-CoV-2 upper respiratory (NP or nasal) swab PCR on the day of inoculation, may be enrolled at the discretion of the investigator.
* Recent blood donation (within prior 56 days).
* Recent or scheduled receipt of any live vaccine 30 days and/or inactivated or sub-unit vaccine 14 days prior to inoculation.
* Safety labs may be repeated once. If outside the 90-day screening window, the volunteer may be rescreened except for flavivirus, hepatitis, and HIV viral screens.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Main/Low Dose DHIM-4: Received 95 pfu DENV-4, primary
- Homologous Rechallenge: Received 95 pfu DENV-4, secondary
Period: Overall Study
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Started | 14 | 6
Detectable DENV Viremia | 14 | 0
Completed | 14 | 5
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.6 [20 to 48] | 32.5 [25 to 48] | 33 [20 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 12 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 8 | 4 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection Site Adverse Events
Description: solicited injection site adverse events until 7 days post virus inoculation
Time Frame: Days 1-7 post-challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants | 1 | 0

2. Primary Outcome: Number of Participants With Unsolicited Injection Site Adverse Events
Description: unsolicited injection site adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: solicited systemic adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants
  Fever | 3 | 0
  Headache/Eye Pain | 10 | 2
  Abdominal Pain | 3 | 0
  Muscle Pain | 9 | 1
  Joint or Bone Pain | 9 | 0
  Fatigue | 14 | 2
  Nausea/Vomiting | 6 | 0
  Rash | 14 | 0

4. Primary Outcome: Incidence of Abnormal Laboratory Measurements
Description: Incidence of abnormal laboratory measurements until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants
  Increased AST (Aspartate Aminotransferase) | 9 | 2
  Increased ALT (Alanine Aminotransferase) | 3 | 2
  Low fibrinogen | 2 | 1
  Leukopenia | 4 | 0
  Neutropenia | 5 | 3
  Low hemoglobin | 4 | 4
  Low glucose | 1 | 0
  High glucose | 1 | 0

5. Primary Outcome: Number of Participants With Dengue-Related Adverse Events
Description: dengue-related like adverse events until 28 days post virus inoculation or 7 days post inpatient whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants
  Fever | 3 | 0
  Headache/Eye Pain | 10 | 2
  Abdominal Pain | 3 | 0
  Muscle Pain | 9 | 1
  Joint/Bone Pain | 9 | 0
  Fatigue | 14 | 2
  Nausea/Vomiting | 6 | 0
  Rash | 14 | 0
  Leukopenia | 4 | 0
  Liver Function Abnormality | 9 | 2
  Thrombocytopenia | 0 | 0

6. Primary Outcome: Number of Participants With Unsolicited Systemic Adverse Events
Description: unsolicited systemic adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants
  Bradycardia | 1 | 0
  Tachycardia | 4 | 2
  Hypertension | 2 | 2
  COVID-19 Infection | 3 | 0
  Nasopharyngitis | 1 | 0
  Pruritis | 2 | 0
  Sensitive Skin | 2 | 0
  Chills | 1 | 0
  Feeling Abnormal | 1 | 0
  Pain | 1 | 0
  Dyspnea | 1 | 0
  Nasal Congestion | 1 | 0
  Oropharyngeal Pain | 1 | 0
  Decreased Appetite | 2 | 0
  Food Poisoning | 0 | 1
  Craniocerebral Injury | 0 | 1

7. Primary Outcome: Number of Participants With Short-Term SAEs
Description: Number of SAEs until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 28
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Long-Term SAEs
Description: Number of SAEs until 6 months post virus inoculation
Time Frame: Days 2, 4-16, 28, 180
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants | 0 | 1

9. Primary Outcome: Number of Participants With Fever
Description: The occurrence of fever defined as greater than or equal to 38°C (100.4° F) measured at least 2 times at least 4 hours apart
Time Frame: Days 2, 4-16, 28, 180
Measure: Count of Participants; unit: Participants
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
Participants | 3 | 0

10. Secondary Outcome: Number of Participants With Detected Viremia
Description: RNAemia measurement by PCR through Day 28 post-challenge. RNA detection is in Cycle threshold (Ct). Viremia is determined by the presence of dengue virus RNA through Day 28 post-challenge. (Was viremia detected?)
Time Frame: Days 2, 4-16, 28
Measure: Number; unit: participants with detected viremia
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
participants with detected viremia | 14 | 0

11. Secondary Outcome: Microneutrilization (50%) Geometric Mean Titer
Description: Microneutrilization (50%) Geometric Mean Titer Dengue antibodies
Time Frame: Day 28
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
Number analyzed (Participants) | 14 | 6
titer | 539.52 [318.64 to 913.49] | 903.69 [284.5 to 2870.54]

ADVERSE EVENTS:
Time Frame: Local Solicited and Unsolicited AEs were quantified through Day 7 post-challenge. Systemic Solicited and Unsolicited AEs were quantified through Day 28 post-challenge. Severe Adverse Events were quantified through 6 months post-challenge.
Arm/Group | Main/Low Dose DHIM-4 | Homologous Rechallenge
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/6
Other Adverse Events (participants affected / at risk) | 14/14 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main/Low Dose DHIM-4 (N=14) | Homologous Rechallenge (N=6)
Injury/Craniocerebral Injury/Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Prior to Day 56 follow-up visit, the participant experienced a traumatic fall from an elevated stairway. Despite ICU measures, the participant succumbed to traumatic brain injury.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main/Low Dose DHIM-4 (N=14) | Homologous Rechallenge (N=6)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (5) | 2 (3)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sensitive Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Feeling Abnormal (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever (Immune system disorders) | 3 | 0
Headache/Eye Pain (General disorders) | 10 | 2
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Muscle Pain (Musculoskeletal and connective tissue disorders) | 9 | 1
Joint or Bone Pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Fatigue (Nervous system disorders) | 14 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 0
Liver Function Abnormality (Hepatobiliary disorders) | 9 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT05268302/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05268302/SAP_001.pdf